CLINICAL TRIAL: NCT05372211
Title: Clinical Use of Recombinant Human Erythropoietin in VLBW and ELBW Infants: a National Survey in China
Brief Title: Survey on the Clinical Use of Recombinant Human Erythropoietin in VLBW and ELBW Infants
Acronym: NSEPO
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shenzhen People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Shenzhen NICUs
Record Dates: First submitted 2022-05-09; First posted 2022-05-12 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2022-05

CONDITIONS: Erythropoietin; Infant; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- General hospital group: Questionnaires collected from general hospitals in China
  Interventions: Other: not use of any intervention
- Maternity and infant hospital group: Questionnaires collected from Maternity and infant hospitals in China
  Interventions: Other: not use of any intervention
- Children's hospital: Questionnaires collected from Children's hospitals in China
  Interventions: Other: not use of any intervention

INTERVENTIONS:
Other: not use of any intervention — not use of any intervention

SUMMARY:
Recombinant human erythropoietin (rhEPO) has been shown to effectively and safely prevent the anemia of prematurity and to reduce the transfusion need in very low birth weight (VLBW) and extremly low birth weight (ELBW) infants and has been licensed for this indication in Europe in 1997. The objective of the study was to obtain information on the use or nonuse of rhEPO in neonatal units in China.

DETAILED DESCRIPTION:
The survey was developed by a team of neonatologists at Shenzhen People's hospital . The survey consisted of 26 questions covering three areas: the characteristics of the survey respondents, the use of rhEPO in VLBW and ELBW infants , and other related questions. The questionnaire was presented in the Questionnaire Star format (https://www.wjx.cn/, Hangzhou Oway Medical Technology,Changsha, China). we plan to conduct a cross-sectional survey through the Neonatal Professional Committee of the Chinese Medical Doctor Association WeChat platform. The questionnaire is going to be distributed to nearly 500 representative neonatologists and pediatricians from general hospitals, maternity and infant hospitals, and children's hospitals across the country. Furthermore, this study was approved by the ethics committee of the Shenzhen People's Hospital.

ELIGIBILITY:
Inclusion Criteria:

neonatologists and pediatricians from general hospitals, maternity and infant hospitals, and children's hospitals across China

Exclusion Criteria:

neonatologists and pediatricians from same hospitals

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Neonatologists and pediatricians from general hospitals, maternity and infant hospitals, and children's hospitals across China
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
The survey (the clinical use of rhEPO) | 01-june-2022
  the clinical use of rhEPO in VLBW and ELBW infants

IPD SHARING:
Plan to Share IPD: Undecided